CLINICAL TRIAL: NCT00936364
Title: Short-Term Fasting Prior To Platinum-based Chemotherapy: Feasibility and Impact on Toxicity
Brief Title: Short-Term Fasting: Impact on Toxicity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0S-08-9
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Fasting in Malignant Solid Tumors
MeSH Terms: interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Stage I of study) (Experimental): Patients fast for 24 hours on day -1
  Interventions: Other: Short-term fasting; Other: Fasting
- Group II (Stage I of study) (Experimental): Patients fast for 48 hours on days -2 and -1
  Interventions: Other: Short-term fasting; Other: Fasting
- Group III (Stage I of study) (Experimental): Patients fast for 72 hours on days -3, -2, and -1
  Interventions: Other: Short-term fasting; Other: Fasting
- Group IV (Stage I of study) (Experimental): Patients undergo a modified 48-hour fast with minimal caloric intake on day -2 and -1
  Interventions: Other: Modified fast; Other: Fasting

INTERVENTIONS:
Other: Short-term fasting — No calories will be consumed during periods of fasting. Good oral hydration will be encouraged. Water may be consumed, as well as non-caloric beverages (i.e. zero calorie soft drinks, black coffee or tea).
  Other Names: fasting
  Arms: Group I (Stage I of study); Group II (Stage I of study); Group III (Stage I of study)
Other: Modified fast — Minimal caloric intake on days -2 and -1
  Other Names: fasting
  Arms: Group IV (Stage I of study)
Other: Fasting — Day -1
  Arms: Group I (Stage I of study)
Other: Fasting — Days -2 and -1
  Arms: Group II (Stage I of study)
Other: Fasting — Days -3, -2, and -1
  Arms: Group III (Stage I of study)
Other: Fasting — 48-hour fast with minimal caloric intake on days -2 and -1
  Arms: Group IV (Stage I of study)

SUMMARY:
This partially randomized clinical trial studies short-term fasting in reducing side effects in patients receiving gemcitabine hydrochloride and cisplatin for advanced solid tumors. Short-term fasting before chemotherapy may reduce the side effects caused by chemotherapy. Drugs used in chemotherapy, such as gemcitabine hydrochloride and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the safety and feasibility of short-term fasting prior to administration of combination chemotherapy with platinum in patients with advanced solid tumor malignancies.

II. To evaluate the toxicity profile of platinum-based chemotherapy in subjects who eat normally compared to those who undertake short-term starvation.

III. To investigate changes in plasma insulin, glucose, IGF1 and IGF binding protein (IGFBP) levels, and oxidative stress markers in subjects who undertake short-term fasting compared to controls.

IV. To investigate whether changes in grp78 expression occur after fasting and after chemotherapy administration in human subjects.

OUTLINE:

STAGE I: Patients are assigned to 1 of 4 treatment groups. GROUP I: Patients fast for 24 hours on day-1.

GROUP II: Patients fast for 48 hours on days -2 and -1.

GROUP III: Patients fast for 72 hours on days -3, -2, and-1.

GROUP IV: Patients undergo a modified 48-hour fast with minimal caloric intake on days -2 and -1.

STAGE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients fast for 72 hours on days -2, and on day 1.

ARM II: Patients proceed to chemotherapy without fasting.

All patients receive gemcitabine hydrochloride intravenously (IV) on days 1 and 8 and cisplatin IV over 2 hours on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confirmed malignancy for which platinum-based chemotherapy on a 21 day cycle or 14 day cycle is being recommended.
* Disease state:

  * Stage I of the trial: newly diagnosed disease for which neoadjuvant or adjuvant chemotherapy is planned in the curative setting, or metastatic disease.
  * Stage II of the trial: Measurable disease by RECIST criteria must be present for all subjects in the randomized component of the trial- if surgery or radiation is planned, the target lesions may not be so treated until after the assessment of the effect of chemotherapy.
* Prior chemotherapy

  * Stage I: subjects may have already received no more than 2 cycle of platinum-based chemotherapy, but should not have received other prior chemotherapy regimens with the exception of patients with metastatic disease who received neoadjuvant or adjuvant chemotherapy and that chemotherapy was completed > 6 months prior to enrollment.
  * Stage II: subjects must have received no prior chemotherapy regimens for metastatic disease, and no more than 2 cycles of their current platinum chemotherapy regimen for metastatic disease. They may have received prior neoadjuvant or adjuvant chemotherapy, provided such therapy was completed >6 months prior to enrollment.
* Prior Radiotherapy is allowed, provided at least 2 weeks have elapsed from completion of radiotherapy to initiation of protocol treatment.
* BMI > 18.5
* ECOG performance status 0-1
* Adequate renal function (Creatinine <1.25 ULIN or calculated creatinine clearance > 50 ml/min)
* Premenopausal women must have a negative pregnancy test and must agree to use barrier contraception throughout the study period.

Exclusion Criteria:

* Diabetes Mellitus
* Recent significant or unexplained weight loss that the investigator feels may pose an unacceptable risk for enrollment. Candidates who are overweight and have lost weight intentionally via diet or exercise should not be excluded.
* Peripheral Neuropathy > grade 1
* History of significant cardiac disease, particularly uncompensated congestive heart failure NYHA grade 2 or more or LVEF < 40% on any prior assessment. (Assessment of LVEF prior to therapy is not required in the absence of other clinical indicators of heart disease). Patients with a prior LVEF <40% will require re-evaluation prior to study entry.
* Subjects on medications that may not be safely stopped during the fasting portion of the study, or which may not be safely consumed without food.
* A history of syncope with calorie restriction in the past or other medical comorbidity, which would make fasting potentially dangerous.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-07-09 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Identification of the longest duration of fasting which is safe | Up to 5 years

SECONDARY OUTCOMES:
Significant toxicity as assessed by CTCAE v3.0 | Up to 5 years
Changes in plasma insulin, glucose, IGF1 and IGF binding protein (IGFBP) levels, and GRP78 expression in WBCs | Up to 2 courses
Changes in grp78 expression after fasting and after chemotherapy administration | After 2 courses

CONTACTS AND LOCATIONS:
Overall Officials: David I Quinn, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehenseive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Dorff TB, Groshen S, Garcia A, Shah M, Tsao-Wei D, Pham H, Cheng CW, Brandhorst S, Cohen P, Wei M, Longo V, Quinn DI. Safety and feasibility of fasting in combination with platinum-based chemotherapy. BMC Cancer. 2016 Jun 10;16:360. doi: 10.1186/s12885-016-2370-6. PMID 27282289